CLINICAL TRIAL: NCT02068014
Title: Implication and Factors Influencing the Decision to Select Srapplers During Laparoscopic Sleeve Gastrectomy.
Brief Title: Standarization for Stappler Application During Sleeve Gastrectomy
Acronym: LSG
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, MD, Assuta Medical Center
Other Study IDs: SA012014
Record Dates: First submitted 2014-02-19; First posted 2014-02-20 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: stapplers- obesity- stomach
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Sleev gastrectomy is a procedure performed for permanent treatment of obesity. For the procedure, cutting of the stomach is performed with differents long of stapplers.

The aim of the study is to determine wich long of stappler is applicable in any stage of the procedure ans the variation expected.

DETAILED DESCRIPTION:
After permormed laparoscopic sleeve gastrectomy the stonach retrieved for pathology study will be messured in three ponts: antrum, body and fundus.

In each point medition of the two walls and any wall (anterior and posterior) will be messurd.

Those data will be stariscally analized to perform a applicable guidelines for stapller selection.

ELIGIBILITY:
Inclusion Criteria:

* every laparoscopic sleeve gastrectomy
* between 18 y.o. and 70 y.o.
* no previous gastric operation

Exclusion Criteria:

* under 18 y.o. or over 70 y.o. previous gastric surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients underwnt laparoscopic sleev gastrectomy between 18 y.o. and 70 y.o.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
differences in wall mesurments | 3 month
  during 3 month the data will be collected and proceceed

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta MC, Tel Aviv, Israel